CLINICAL TRIAL: NCT07010770
Title: SMART Therapist Training: A Hybrid Factorial-SMART Design
Acronym: SMART
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: IIR 24-069; HX003943-01 (Other Grant/Funding Number: VA HSRD)
Record Dates: First submitted 2025-05-30; First posted 2025-06-08 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Stress Disorders, Post-Traumatic; Psychotherapy
Keywords: Therapeutics; Psychotherapy; Stress Disorders, Post-Traumatic; Referral and Consultation; Veterans
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: All eligible participants will initially be randomized to one of the first-stage tactics:
  1. Web-Based Training (WBT) + Consultation with Work-Sample Review (WR)
  2. Web-Based Training (WBT) + Standard Consultation
  3. Standard Training + Consultation with Work-Sample Review (WR)
  4. Standard Training + Standard Consultation
  After four months/one completed case, CPT fidelity will be assessed, and therapists who demonstrate inadequate fidelity/cannot be reached for assessment will be classified as demonstrating "fidelity in progress" and will be re-randomized to one of two second-stage tactics for the next two months:
  1. Continue in standard consultation
  2. Step up to high intensity consultation with biweekly session review.
     Therapists who have achieved fidelity benchmarks will be classified as demonstrating "early fidelity" and will be re-randomized to one of two second-stage tactics for the next two months:
  3. Continue in standard consultation
  4. Step down to fidelity self-monitoring
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (16):
- Condition 1-A (Experimental): Web-Based Training (WBT) + Work-Sample Review (WR) + early fidelity + step down to fidelity self-monitoring.
  Interventions: Other: Web-Based Training (WBT); Other: Work Sample Review (WR); Other: Step down to fidelity self-monitoring
- Condition 1-B (Experimental): Web-Based Training (WBT) + Work-Sample Review (WR) + early fidelity + continue in Standard Consultation.
  Interventions: Other: Web-Based Training (WBT); Other: Work Sample Review (WR)
- Condition 1-C (Experimental): Web-Based Training (WBT) + Work-Sample Review (WR) + fidelity in progress + step up to session audio review.
  Interventions: Other: Web-Based Training (WBT); Other: Work Sample Review (WR); Other: Step up to session audio review
- Condition 1-D (Experimental): Web-Based Training (WBT) + Work-Sample Review (WR)+ fidelity in progress + continue in Standard Consultation.
  Interventions: Other: Web-Based Training (WBT); Other: Work Sample Review (WR); Other: Continue in Standard Consultation
- Condition 2-A (Experimental): Web-Based Training (WBT) + Standard Consultation (SC) + early fidelity + step down to fidelity self-monitoring.
  Interventions: Other: Web-Based Training (WBT); Other: Step down to fidelity self-monitoring; Other: Standard Consultation (SC)
- Condition 2-B (Experimental): Web-Based Training (WBT) + Standard Consultation (SC) + early fidelity + continue in Standard Consultation.
  Interventions: Other: Web-Based Training (WBT); Other: Standard Consultation (SC)
- Condition 2-C (Experimental): Web-Based Training (WBT) + Standard Consultation (SC) + fidelity in progress + step up to session audio review.
  Interventions: Other: Web-Based Training (WBT); Other: Step up to session audio review; Other: Standard Consultation (SC)
- Condition 2-D (Experimental): Web-Based Training (WBT) + Standard Consultation (SC) + fidelity in progress + continue in Standard Consultation.
  Interventions: Other: Web-Based Training (WBT); Other: Standard Consultation (SC); Other: Continue in Standard Consultation
- Condition 3-A (Experimental): Standard Training (ST) + Work-Sample Review (WR) + early fidelity + step down to fidelity self-monitoring.
  Interventions: Other: Work Sample Review (WR); Other: Step down to fidelity self-monitoring; Other: Standard Training (ST)
- Condition 3-B (Experimental): Standard Training (ST) + Work-Sample Review (WR) + early fidelity + continue in Standard Consultation.
  Interventions: Other: Work Sample Review (WR); Other: Standard Training (ST)
- Condition 3-C (Experimental): Standard Training (ST) + Work-Sample Review (WR) + fidelity in progress + step up to session audio review.
  Interventions: Other: Work Sample Review (WR); Other: Step up to session audio review; Other: Standard Training (ST)
- Condition 3-D (Experimental): Standard Training (ST) + Work-Sample Review (WR)+ fidelity in progress + continue in Standard Consultation.
  Interventions: Other: Work Sample Review (WR); Other: Standard Training (ST); Other: Continue in Standard Consultation
- Condition 4-A (Experimental): Standard Training (ST) + Standard Consultation (SC) + early fidelity + step down to fidelity self-monitoring.
  Interventions: Other: Step down to fidelity self-monitoring; Other: Standard Consultation (SC); Other: Standard Training (ST)
- Condition 4-B (Experimental): Standard Training (ST) + Standard Consultation (SC) + early fidelity + continue in Standard Consultation.
  Interventions: Other: Standard Consultation (SC); Other: Standard Training (ST); Other: Continue in Standard Consultation
- Condition 4-C (Experimental): Standard Training (ST) + Standard Consultation (SC) + fidelity in progress + step up to session audio review.
  Interventions: Other: Step up to session audio review; Other: Standard Consultation (SC); Other: Standard Training (ST)
- Condition 4-D (Experimental): Standard Training (ST) + Standard Consultation (SC) + fidelity in progress + continue in Standard Consultation.
  Interventions: Other: Standard Consultation (SC); Other: Standard Training (ST); Other: Continue in Standard Consultation

INTERVENTIONS:
Other: Web-Based Training (WBT) — A self-paced online training course that includes video demonstrations, self-guided modules, and clinical materials/resources.
  Arms: Condition 1-A; Condition 1-B; Condition 1-C; Condition 1-D; Condition 2-A; Condition 2-B; Condition 2-C; Condition 2-D
Other: Work Sample Review (WR) — Four months of weekly hour-long consultation that will include trainer-led reviews of work samples, focusing on the Impact Statement and Stuck Point Log.
  Arms: Condition 1-A; Condition 1-B; Condition 1-C; Condition 1-D; Condition 3-A; Condition 3-B; Condition 3-C; Condition 3-D
Other: Step down to fidelity self-monitoring — After four months, and for participants who are classified as meeting "early fidelity", for the next two months, therapists in self-monitored fidelity will no longer attend group consultation. Instead, they will assess their own fidelity through self-report surveys.
  Arms: Condition 1-A; Condition 2-A; Condition 3-A; Condition 4-A
Other: Step up to session audio review — After four months, and for participants who are classified as meeting "fidelity in progress", for the next two months, therapists will have their session audio recordings reviewed and rated for fidelity.
  Arms: Condition 1-C; Condition 2-C; Condition 3-C; Condition 4-C
Other: Standard Consultation (SC) — Four months of weekly hour-long group consultation
  Arms: Condition 2-A; Condition 2-B; Condition 2-C; Condition 2-D; Condition 4-A; Condition 4-B; Condition 4-C; Condition 4-D
Other: Standard Training (ST) — 2-day instructor-led CPT workshop.
  Arms: Condition 3-A; Condition 3-B; Condition 3-C; Condition 3-D; Condition 4-A; Condition 4-B; Condition 4-C; Condition 4-D
Other: Continue in Standard Consultation — After four months, therapists will continue to attend weekly hour-long group consultation for another two months.
  Arms: Condition 1-D; Condition 2-D; Condition 3-D; Condition 4-B; Condition 4-D

SUMMARY:
Cognitive Processing Therapy (CPT) is highly effective in randomized controlled trials, but its effectiveness drops substantially in standard clinical practice, largely due to therapist "drift" from fidelity to the protocol. What remains unknown is which components of CPT training yield high therapist fidelity. Thus, there is a critical need to use empirical approaches to identify the most effective components of CPT training and to develop an adaptive training model for CPT by testing sequences of empirically-supported training strategies. The long-term goal of this research is to develop a sustainable model of therapy training that is personalized to the needs of the therapist trainee.

The overall objective of this application is to empirically optimize an adaptive model for CPT training. The rationale is that developing an adaptive training model will improve efficiency and personalization, yield higher fidelity, and ultimately improve Veteran outcomes. We expect that completion of this project will produce an adaptive CPT training program that yields high therapist fidelity. Improving CPT fidelity in VHA will have a positive impact on the health and wellbeing of Veterans with PTSD.

DETAILED DESCRIPTION:
Background: One third of post-9/11 Veterans in VHA suffer from posttraumatic stress disorder (PTSD), and even among those who receive evidence-based PTSD treatment, over half remain symptomatic. Cognitive Processing Therapy (CPT) is a first-line treatment for PTSD that is initiated three times more frequently than any other trauma-focused treatment. CPT is highly effective in randomized controlled trials, but its effectiveness drops substantially in standard clinical practice, largely due to therapist "drift" from fidelity to the protocol. What remains unknown is which components of CPT training yield high therapist fidelity. Thus, there is a critical need to use empirical approaches to identify the most effective components of CPT training and to develop an adaptive training model for CPT by testing sequences of empirically- supported training strategies. The long-term goal of this research is to develop a sustainable model of therapy training that is personalized to the needs of the therapist trainee. The overall objective of this application is to empirically optimize an adaptive model for CPT training. The rationale is that developing an adaptive training model will improve efficiency and personalization, yield higher fidelity, and ultimately improve Veteran outcomes. We expect that completion of this project will produce an adaptive CPT training program that yields high therapist fidelity. Improving CPT fidelity in VHA will have a positive impact on the health and wellbeing of Veterans with PTSD.

Significance: The number of VHA patients with a diagnosis of PTSD has steadily increased for the past 10 years, therefore improving VHA's capacity to deliver PTSD treatment is of utmost importance. This project aligns with the 2024 VHA priorities to connect Veterans to the best care and improve VHA workforce retention.

Innovation & Impact: Upon successful completion of this project, we expect to contribute an empirically-based, adaptive training model for CPT. This contribution will improve therapist fidelity to CPT and ultimately yield superior clinical outcomes for Veterans with PTSD. The research is innovative because it will use a novel, highly efficient experimental design to shift the current CPT training paradigm from fixed, hard-to-scale strategies to a dynamic and accessible approach, composed of empirically-based components. Our specific aims are:

* Specific Aim 1: Identify which of two low-intensity training components contribute meaningfully to therapist fidelity. We will test the effectiveness of each component and their interaction, as measured by therapist fidelity ratings across 12 months.
* Specific Aim 2: For those with "fidelity in progress," determine whether stepping up to high-intensity consultation improves fidelity. We hypothesize that stepping up will lead to greater fidelity.
* Exploratory Aims: A) For those with "early fidelity," assess the impact of stepping down to self-monitoring versus continuing in standard consultation. B) Compare standard training and consultation to the embedded adaptive training strategies. C) Identify moderators. D) Conduct cost analysis and refine the program through process evaluation.

Methodology: This Hybrid Factorial-SMART will determine which of two low-intensity components (Web-based Training or Consultation Work-Sample Review) is most effective during the initial phase of CPT training. Those who have reached fidelity benchmarks at Month 4 ("early fidelity") will be re-randomized to Continue with standard consultation or Step Down to fidelity self-monitoring. Those not reaching fidelity at Month 4 ("fidelity in progress") will be re- randomized to Continue or Step Up to high-intensity consultation. Fidelity will be assessed by trained evaluators at baseline, 6, 9, & 12 months via standardized patient exercise.

ELIGIBILITY:
Inclusion Criteria:

We have designed the sample to be representative of therapists who are eligible for CPT rollout training.

* Participants must be licensed mental health clinicians or a mental health trainee in VA service (e.g., practicum students, psychology interns, postdoctoral fellows) whose formal job responsibilities include the provision of psychotherapy services to Veterans on a regular basis
* Participants must be able to participate for 9 months.
* Participants must work in a setting where CPT may be implemented (12 weekly 60-minute individual sessions or 90-minute group sessions).
* Participants must have local/supervisor support to implement CPT and fully participate in all training and consultation activities.
* Participating trainees (e.g. psychology interns) on a 6-month training rotation must have permission from their supervisors to continue the study into their next rotation.

Exclusion Criteria:

* Participant is not a licensed mental health clinician
* Participant is already certified in CPT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2030-05-31 (Estimated); Study Completion 2030-08-30 (Estimated)

PRIMARY OUTCOMES:
CPT Therapist Adherence and Competence Scale (TAC) | Baseline (0-months), 6-months, 9-months, and 12-months.
  The TAC measures both adherence to specific unique and essential CPT elements, and competence in delivering these interventions.
  Adherence is rated on a 3-point Likert-type scale, with 0=incomplete, 1=mostly complete, and 2=fully complete as prescribed in each session.
  Competence is rated on a 7-point Likert-type scale, from 0=not competent to 6=outstanding competence. Items rated as a "0" on adherence are automatically rated a "0" for competence. Competence scores between 0 and 2 are cases in which the therapist requires "substantial corrective feedback." Scores between 3 and 4 indicate "acceptable to good; opportunities for feedback," such that the therapist performs the intervention well, but has room for improvement. Scores of 5 and 6 require very little to no feedback.

SECONDARY OUTCOMES:
The Cognitive Therapy Scale-Revised (CTS-R) | Baseline (0-months), 6-months, 9-months, and 12-months.
  The CTS-R assesses transdiagnostic CBT specific skills (Guided discovery, Conceptualization, Identifying key cognitions, Application of change methods, Application of behavioral techniques, Homework, and Facilitation of emotional expression) and general therapeutic skills (Agenda, Feedback, Collaboration, Pacing/use of time, and Interpersonal effectiveness). Items are rated on a 0 = incompetent (non-compliance) to 6 = expert (compliance + high skill) scale with item-specific descriptions for each anchor. The range of scores is 0-72.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Kaufman Sripada, PhD MS, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI
Locations (4):
- United States (4):
  - VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California
  - VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan
  - Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota
  - Cincinnati VA Medical Center, Cincinnati, OH, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No